CLINICAL TRIAL: NCT06440460
Title: Social and Biological Mechanisms Driving the Intergenerational Impact of War on Child Mental Health: Implications for Developing Family-Based Interventions
Brief Title: Intergenerational Study of War-Affected Youth
Acronym: ISWAY
Status: Active, not recruiting | Type: Observational
Sponsor: Boston College (Other)
Collaborators: University of Makeni (Unknown); Caritas Freetown (Other); Tulane University (Other); Kenema Government Hospital (Other)
Responsible Party: Principal Investigator, Theresa Betancourt, Salem Professor in Global Practice, Boston College
Other Study IDs: 22.115.01
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorders; Anxiety State; Depressive Disorder; Mood Disorders; Trauma and Stressor Related Disorders; Social Skills; Violence, Non-accidental
Keywords: Early Child Development; Sierra Leone; Observational Study; Longitudinal; Emotion Regulation; Self Regulation; Mental Health; Stress; Trauma; Quality of Life; Stress Biomarkers; Biological Embedding; Parenting
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Mood Disorders; Trauma and Stressor Related Disorders; Social Skills; Emotional Regulation; Self-Control; Psychological Well-Being; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
War-related violence is a leading driver of mental disorders and illness affecting children in low- and middle-income countries (LMICs). Parents exposed early in life to war-related violence and loss are at risk for mental health problems and may pass risks to their offspring. The study posits that war-related trauma alters the stress-response circuitry in ways that endure into adulthood and affect the next generation. This will be the first investigation in a 20-year longitudinal study to examine mechanisms that link parental war-related trauma exposure and subsequent mental health problems to risk for mental disorders in offspring. This study will extend the first intergenerational study of war in Sub-Saharan Africa (R01HD073349) to focus on children (aged 7-24) born to war-affected parents. Assessments of behavioral and biological indicators of the Research Domain Criteria (RDoC)-linked constructs of self-regulation and stress reactivity will be collected, including autonomic nervous system reactivity, inflammation, and telomere length as well as sophisticated observations of parent-child interactions and synchrony. These measures will be utilized to identify potentially modifiable risk and protective processes both to inform the development of screening tools to identify families at risk for poor child mental health and to be deployed as active ingredients of interventions to reduce transmission of mental health problems to children of war-affected parents.

This follow-up study involves the following activities:

1. Pilot to assess measure performance and field test study protocols.

   1. Translation and adaptation of newly selected measures
   2. Pilot study of new child and adult measures with 36 caregivers and 60 children in a district of Sierra Leone unlinked to participants to test the feasibility and validity of new tools.
2. Fifth wave of data collection from war-affected youth who are now parents and their children aged 7-24.

   1. Household tracking and re-enrollment of 145 households that were formerly enrolled in the Longitudinal Study of War-Affected Youth (LSWAY; T1: 2002, T2: 2004, T3: 2008, T4: 2016).
   2. Quantitative (full sample) and qualitative (subsample) data collection with 145 households who were enrolled in T4 LSWAY, including war-affected youth who are now parents, their intimate partners, and their children aged 7-24.

Through these activities, the investigators will test three overarching hypotheses:

1. Childhood war-related trauma exposure will be associated with mental difficulties (anxiety, depression, post-traumatic stress, disruptions of emotion regulation).
2. Poor mental health in war-affected parents will be associated with emotional and behavioral disruptions in biological offspring.
3. Risk and protective factors across the social ecology may serve as intervention targets to mitigate the effects of parental war-related trauma on behavioral disruptions and stress physiology, both within and across generations.

DETAILED DESCRIPTION:
The Intergenerational Study of War-Affected Youth (ISWAY) entails a fifth wave of data collection in a 22-year study of war-affected youth in Sierra Leone (LSWAY), the first of its kind in Sub-Saharan Africa. LSWAY findings drawn from four waves of data collection (T1:2002, T2: 2004, T3: 2008, T4:2016/17) indicate that a healthy transition to adulthood among war-affected youth was linked to engagement in prosocial behavior and community involvement, while problems with hostility, poor emotion regulation, and social withdrawal created barriers to achieving healthy and productive lives. Community stigma and poor family acceptance compounded these barriers. Preliminary analyses of offspring of war-affected youth-first enrolled at T4-indicated that harsh paternal parenting was associated with offspring poor mental health and maternal parenting (harsh and warm) predicted offspring disruptions in emotion regulation and mental health. The investigators theorize such associations are linked to biological mechanisms, but research to date has been limited to cross-sectional data on the health and mental health of biological offspring.

ISWAY will examine how social and biobehavioral mechanisms operate among war-affected parents to shape parenting and the mental health of offspring. The study's guiding framework blends a biobehavioral and ecological model of risk and resilience with the Stress Adjustment Paradigm.The Multisystemic Model of Child Development holds that both behavioral and biological mechanisms are influenced by risk and protective factors at different levels of the social ecology and that exposure to trauma may lead to disruptions in individual stress reactivity and emotion regulation. The Stress-Adjustment Paradigm posits that traumatic life events lead to individual outcomes that are shaped by risk and protective processes across the social ecology. Taken together, these theories propose that both past trauma and current social stressors (e.g., underemployment, stigma) have implications for understanding the mechanisms linking past parental trauma to parent-child interactions and the mental health of subsequent generations. Adult stress reactivity, including ANS reactivity, may manifest in similar ways among offspring. Biological markers of inflammation and telomere length may also be linked in war-affected parents and their offspring. An integrated model suggests that several important protective processes and resources may operate to mitigate these intergenerational disruptions such as social support and access to other attachment figures in the household who have strong self-regulation. Helping parents who have experienced severe trauma build self-regulation skills and extending social support networks may be critical components of preventive interventions.

ISWAY entails an enriched follow-up of the parents and their offspring focusing on the RDoC-related constructs that may underlie self-regulation (negative/positive valence systems, arousal systems, social processes). Collecting and analyzing both behavioral and biological/physiological data will deepen understanding of mechanisms that may contribute to increased risk of mental health difficulties in offspring. This will be amplified by an exploration of modifiable risk and protective factors across the social ecology (individual, family, and community levels) to prioritize as intervention targets for addressing intergenerational risks to the mental health of offspring of war-affected parents.

ELIGIBILITY:
Inclusion Criteria:

* being a war-affected young adult (referred to as the index participant) previously interviewed at one or more waves of the Longitudinal Study of War Affected Youth (LSWAY) who still resides in Sierra Leone
* being a cohabitating intimate partner of the index participant; or (c) being a cohabitating biological child (aged 7-24) of the index participant. Exclusion criteria are (a) not being sampled in a prior LSWAY wave
* being a cohabitating biological child (aged 7-24) of the index participant

Exclusion Criteria:

* not being sampled in a prior LSWAY wave
* not being a biological child or intimate partner of the index cohort participant
* being in acute crisis (active suicidality or psychosis)

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of participants who were formerly enrolled in T4 of LSWAY, including index subjects (i.e., war-affected youth), their caregivers, and biological offspring who meet the eligibility criteria. In addition, focus group participants, who were not part of the LSWAY cohort from prior study waves, will be recruited from the 5 largest districts in which LSWAY participants reside. These participants will be sampled in order to understand community experiences regarding the social context of parenting in Sierra Leone, including challenges and perceptions of social norms and their effect on everyday life in Sierra Leone.
Sampling Method: Non-Probability Sample
Enrollment: 804 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist (HSCL) | May-December 2024
  The HSCL is a diagnostic tool for depression and anxiety in caregivers and consists of 25 items, including 10 items for anxiety symptoms and 15 items for depression symptoms. Response options are Not at All (1), A Little (2), Quite a Bit (3), and Extremely (4) with higher scores indicating more symptoms.
Center for Epidemiological Studies Depression Scale-Child (CESD-Child) | May-December 2024
  The CESD-Child is a diagnostic tool for depression in children. Caregiver and child self-report versions include 20 items with response options including Never (0), A little (1), Sometimes (2), and Often (A Lot) (3) with higher values indicating more symptoms.
UCLA PTSD Reaction Index-Revised (UCLA PTSD-RI) | May-December 2024
  The UCLA PSTD-RI is a diagnostic tool for post-traumatic stress disorder. An adult self-report version includes 23 items assessing trauma history, scored according to whether the event occurred or not (0 = No, 1 = Yes), and 12 items on PTSD symptoms with response options including Never (0), Sometimes (1), and Often (2) with higher values indicating more symptoms. A child self-report version includes 14 items assessing trauma history, scored according to whether the event occurred or not (0 = No, 1 = Yes), and 11 items on PTSD symptoms with response options including Never (0), Sometimes (1), and Often (2) with higher values indicating more symptoms.
Child Behavior Checklist (CBCL) | May-December 2024
  The CBCL includes child self-report and caregiver report on child's internalizing and/or externalizing behavior. The caregiver report includes 118 items with response options including Not True (0), Somewhat or Sometimes True (1), and Very True or Often True (2). Scores are summed within 8 syndrome scales (Withdrawn, Somatic Complaints, Anxious/Depressed, Social Problems, Thought Problems, Attention Problems, Delinquent Behavior, and Aggressive Behavior) with higher scores indicating more symptoms. The child self-report includes 102 items with the same response options and subscales as the caregiver version. Higher scores indicate more symptoms.
Difficulties in Emotion Regulation Scale (DERS) | May-December 2024
  The DERS includes caregiver self-report and child self-report on emotion regulation. There are 36 items that measure six subscales: nonacceptance of emotional responses; difficulty engaging in goal-directed behavior; impulse control difficulties; lack of emotional awareness; limited access to emotion regulation strategies; lack of emotional clarity. Response options are Almost Never (1), Sometimes (2), About Half the Time (3), Most of the Time (4), and Almost Always (5) with higher scores indicating greater difficulties in emotion regulation.
Oxford Measure of Psychosocial Adjustment (OMPA) | May-December 2024
  The OMPA includes child self-report and caregiver report on child of externalizing, internalizing, and prosocial attitudes and behaviors. The full scale includes 53 items measuring four subscales: anxiety and depression; hostility; pro-social behavior; and confidence. Response options are Never (1), Hardly (2), Sometimes (3), and Always (4) with higher scores indicating more symptoms.
Rapid Assessment of. Cognitive and Emotional Regulation (RACER) | May-December 2024
  Observation of child and caregiver cognitive functioning
Kaufman Assessment Battery for Children | May-December 2024
  Observation of child's
SWAY Parenting | May-December 2024
  The SWAY Parenting scale includes caregiver report on family information such as the number of biological and non-biological children, numbers of children, and history of pregnancy, followed by 15 Likert-scale items that ask about caregiving behaviors (e.g., time spent playing with child, reading to child, telling stories, etc.). Response options are Never (0), Sometimes (1), Often (2), and Always (3) with higher scores indicating more engagement in caregiving behaviors.
Adapted UNICEF Multiple Indicator Cluster Survey Child Discipline Module | May-December 2024
  Caregiver self-report of child discipline practices and behaviors
Parenting Acceptance and Rejection Questionnaire (PARQ) | May-December 2024
  The PARQ Short Form includes caregiver self-report and child report on caregiver versions with 23 items and four subscales (warmth/affection, hostility/aggression, indifference/neglect, and undifferentiated rejection). Response options are Almost Never True (1), Rarely True (2), Sometimes True (3), and Almost Always True (4) with higher scores indicating more frequent behaviors.
Coding Interactive Behavior | May-December 2024
  Coding system for observation of caregiver-child interactions
Early Grade Reading Assessment Early Grade Reading Assessment | May-December 2024
  Observation of child's early literacy skills
Early Grade Math Assessment | May-December 2024
  Observation of child's early numeracy skills
Autonomic Stress Reactivity | May-December 2024
  Measure of caregiver and child's autonomic response to stress via respiratory sinus arrhythmia (RSA)
Telomere Length | May-December 2024
  Measure of caregiver and child's telomere length
Inflammation | May-December 2024
  Measure of caregiver and child's inflammatory markers (e.g., C-reactive protein)
Post-War Adversities Scale | May-December 2024
  The Post-War Adversities Scale is an adult self-report scale that includes 18 items asking about daily hardships within the past three months (e.g., inadequate living accommodations, eviction, serious conflicts, etc) and 11 items asking about daily hardships within the past 12 months (e.g., being robbed, very ill, deaths, financial crisis, etc.). Response options are No (0) and Yes (1). Higher scores indicate more adversities.
Perceived Stress Scale (PSS) | May-December 2024
  The PSS is an adult self-report scale with 10 items asking about perceptions of stressful feelings (e.g., unable to cope, feeling nervous and stressed, being angered, etc.). Response options include Never (0), Almost Never (1), Sometimes (2), Fairly Often (3), and Very Often (4) with higher scores indicating more feelings of distress.
Childhood Trauma Questionnaire (CTQ) | May-December 2024
  The CTQ is an adult self-report scale with five subscales including emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Response options include Never (0), Hardly (1), Sometimes (2), and Always (3) with higher scores indicating more abuse or neglect.

SECONDARY OUTCOMES:
Brief COPE Scale | May-December 2024
  The Brief COPE is an adult self-report scale that includes 14 subscales with two items each for a total of 28 items. Subscales include: self-distraction; active coping; denial; substance use; use of emotional support; use of instrumental support; behavioral disengagement; venting; positive reframing; planning; humor; acceptance; religion; and self-blame. Response options include Not at All (1), A Little (2), Some (3), and A Lot (4) with higher scores indicating more endorsement of the coping style.
Normative Beliefs about Aggression Scale (NBA) | May-December 2024
  The NBA is a 20-item scale that can be used with children, adolescents, and adults to measure perceptions of how acceptable it is to behave aggressively under different conditions. Response options include It's Really Wrong (0), It's Sort of Wrong (1), It's Sort of OK (2), and It's Perfectly OK (3) with higher scores indicating a more accepting disposition toward aggression.
Post-Traumatic Growth Inventory (PTGI) | May-December 2024
  The PTGI is a caregiver self-report scale with 21 items and five subscales including relating to others, new possibilities, personal strength, spiritual change, and appreciation of life. Response options include: I did not experience this change (1), I experienced this change to a very small degree (2), I experienced this change to a small degree (3), I experienced this change to a moderate degree (4), I experienced this change to a great degree (5), and I experienced this change to a very great degree (6). Higher scores indicate more post-traumatic growth.
Adapted Youth Risk Behavior Survey | May-December 2024
  Child and caregiver self-report of risk behaviors
WHO Disability Adjustment Scale (WHODAS) | May-December 2024
  The WHODAS is an adult and child self-report scale that includes 12 items asking about difficulties with functioning within the past 30 days. Response options include None (0), Mild (1), Moderate (2), Severe (3), and Extreme or Can't Do (4) with higher scores indicating more difficulties.
Child Rating Scale (CRS) | May-December 2024
  The CRS is a child self-report scale that includes 40 items and four subscales including rule compliance/acting out, anxiety/withdrawal, interpersonal social skills, and self-confidence. Response options are Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), and Strongly Agree (4) with higher scores indicating more endorsement of the trait.
Demographic and Health Survey (DHS) - Intimate Partner Violence (IPV) | May-December 2024
  The IPV scale is an adult self-report scale of intimate partner violence perpetration and victimization. The scale includes 20 perpetration items and 20 victimization items on emotional, physical, and sexual abuse within the previous three months. Response options are This Has Never Happened (0), Once in the Past Three Months (1), Twice in the Past Three Months (2), 3 to 5 Times in the Past Three Months (3), 6 to 10 Times in the Past Three Months (4), 11-20 times in the Past Three Months (5), More than 20 Times in the Past Three Months (6), Not in the Three Months, but It Did Happen Before (7). The questionnaire is scaled such that higher values indicate more intimate partner violence.
Dyadic Adjustment Scale (DAS) | May-December 2024
  The DAS is an adult self-report measure of relationship quality with 32 items and four subscales including dyadic consensus, dyadic satisfaction, dyadic cohesion, and affectional expression. The scale is scored such that higher scores indicate more positive characteristics within each subscale.
Demographic and Health Survey (DHS) Sierra Leone Household Module | May-December 2024
  Caregiver and adult child report on demographic and household information
Perceived Community Acceptance (PCA) | May-December 2024
  The PCA scale is an adult self-report scale that includes 12 items on perceptions about one's acceptance within the community. Response options are Not True (1), Sometimes/Somewhat True (2), and Very True (3) with higher scores indicating more community acceptance.
Collective Efficacy Scale (CES) | May-December 2024
  The CES is an adult self-report measure of perceptions of cohesion and mutual trust within the community. The scale is scored to measure two dimensions, collective efficacy and community disorder, with higher scores indicating more endorsement of the subscale characteristic.
Everyday Discrimination Scale (EDS) | May-December 2024
  The EDS is an adult self-report measure of interpersonal discrimination that is either chronic or episodic. Response options are Never (0), Sometimes (1), and Always (2) with higher scores indicating more experiences of discrimination.
Inventory of Socially Supportive Behaviors (ISSB) | May-December 2024
  The ISSB is an adult and child self-report measure of social support. The version used in this study is adapted to the local context and consists of 25 Likert-style items asking about whether the participant had relationships with people who provided various kinds of social support within the previous month. Response options include It Never Happened (1), It Happened One or Two Times Per Month (2), It Happened One Time Per Week (3), It Happened Several Times Per Week (4), It Happened Almost Every Day (5), with higher scores indicating more social support.
Gender Equitable Men scale (GEM) | May-December 2024
  The GEM Short Form is an adult scale measuring attitudes about gender roles with 9 items. Response options include Do Not Agree (0), Partially Agree (1), and Agree (2) with higher scores indicating more inequitable beliefs about gender roles.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa S Betancourt, Principal Investigator — Boston College
Locations (1):
- Caritas Freetown, Freetown, Sierra Leone

IPD SHARING:
Plan to Share IPD: No